CLINICAL TRIAL: NCT04229615
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase III Clinical Trial Evaluating the Efficacy and Safety of Fluzoparib±Apatinib for Maintenance Treatment in Patients With Advanced Ovarian Cancer Who Have Achieved Effective Response After First-line Platinum-containing Chemotherapy
Brief Title: A Study of Fluzoparib±Apatinib Versus Placebo Maintenance Treatment in Patients With Advanced Ovarian Cancer Following Response on First-Line Platinum-Based Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FZPL-Ⅲ-302
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — fluzoparib; apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety Lead-in, Doublet Arm (Experimental): Fluzoparib+Apatinib
  Interventions: Drug: Fluzoparib; Apatinib
- Single Arm (Experimental): Fluzoparib
  Interventions: Drug: Fluzoparib
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluzoparib; Apatinib — Drug: Fluzoparib Orally twice daily; Apatinib Orally once daily
  Arms: Safety Lead-in, Doublet Arm
Drug: Fluzoparib — Fluzoparib Orally twice daily
  Arms: Single Arm
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, blinded, 3-arm Phase 3 study to evaluate the efficacy and safety of Fluzoparib alone or with Apatinib versus Placebo, as maintenance treatment, in patients with Stage III or IV ovarian cancer. Patients must have completed first-line platinum based regimen with Complete Response (CR) or Partial Response (PR). The study contains a Safety Lead-in Phase in which the safety and tolerability of Fluzoparib+Apatinib will be assessed prior to the Phase 3 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* （phase 3）Histologically new diagnosed, advanced (FIGO Stage III or IV) high-grade serous or endometrioid ovarian cancer (including primary peritoneal and fallopian tube cancer)
* （phase 3）Complete response (CR) or partial response (PR) achieved with front-line platinum-based chemotherapy regimen as determined by investigator
* （phase 3）Ability to be randomized ≤8 weeks after last dose of platinum
* （Saftey Lead-in）Received 2~4 prior chemotherapy regimens. Platimun sensitive relapsed; Have at least one measurable disease as defined by RECIST v1.1.

Exclusion Criteria:

* Prior treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor or Apatinib
* Patients who have received other study drug treatment within 4 weeks prior to the first administration(< 5 elimination half-lives of the study drug molecular targeted anti-cancer drugs).
* Patients with clinical symptoms of cancer ascites, pleural effusion, who need to drainage, or who have undergone ascites drainage within 2 months prior to the first administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
(Safety Lead-in) Incidence of ≥3 grade TRAEs | up to 28 days after the last patient of the lead-in phase
  Incidence of ≥3 grade treatment related adverse events
(Phase 3) Progression free survival(PFS) in advanced ovarian cancer patients | up to 4 years
  Defined as progression free survival per RECIST 1.1 criteria according to BIRC criteria

SECONDARY OUTCOMES:
AEs+SAEs | from the first drug administration to within 30 days for the last treatment dose
  Adverse Events and Serious Adverse Events
PFS by investigator's assessment | up to 4 years
  Progression-Free-Survival
OS | up to 6 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up
Patients reported outcome（PROs）assessed by EQ-5D-5L questionnaire | 48 months
  Comparison of the Quality of Life in study arms assessed by EQ-5D-5L questionnaire
Patients reported outcome（PROs）assessed by FOSI questionnaire | 48 months
  Comparison of the Quality of Life in study arms assessed by FOSI questionnaire
Time to progression on the next anticancer therapy (PFS2) From date of start of next anticancer therapy to date of first documented progression of date of death from any cause, whichever comes first. | 4 years
  From date of start of next anticancer therapy to date of first documented progression of date of death from any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided